CLINICAL TRIAL: NCT04032834
Title: A Randomized, Open-label, Crossover Trial to Compare the Pharmacokinetics, Safety and Tolerability of Single Doses of VR647 Inhalation Suspension Delivered by the VR647 Inhalation System (VR647) With Single Doses of Budesonide Delivered by a Conventional Jet Nebulizer in Healthy Adult Volunteers and Adult Asthma Subjects
Brief Title: A Comparison of VR647 and Conventionally Nebulized Budesonide in Healthy Volunteers and Adult Asthma Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vectura Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR647/1/001
Record Dates: First submitted 2019-07-04; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Asthma; Budesonide; Nebulizer; Pharmacokinetics; AKITA JET
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: This is a three part, randomized, open-label, crossover, Phase 1 trial in adults. Parts 1 and 2 are comparative single dose, 6-treatment, 6-period crossover trials with a mouthpiece or facemask, respectively, in healthy adults. Subjects will receive 4 dose levels of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (AKITA JET) (5, 10, 15 and 25 breaths, with a targeted doses of 30, 60 120 and 240 µg) and 2 dose levels of budesonide delivered by conventional jet nebulizer (PARI VIOS) (0.5 and 1 mg). Part 3 is a comparative single dose, 4-treatment, 4-period crossover trial in subjects with mild asthma. Subjects will receive doses of VR647 Inhalation Suspension (15 breaths, with a targeted dose of 120 µg) delivered by the VR647 Inhalation System (AKITA JET) with facemask or mouthpiece and budesonide (0.5 mg) delivered by conventional jet nebulizer (PARI VIOS) with facemask or mouthpiece.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Part 1, Arm A of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece
- Part 1, Arm B of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece
- Part 1, Arm C of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece
- Part 1, Arm D of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece
- Part 1, Arm E of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece
- Part 1, Arm F of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece
- Part 2, Arm A of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 2, Arm B of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 2, Arm C of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 2, Arm D of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 2, Arm E of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647, 10 breaths (60 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 2, Arm F of single-dose, 6-treatment, 6-period crossover (Other): Subjects received the following treatments in Periods 1 to 6 in a crossover fashion: 10 breaths (60 µg) VR647, 15 breaths (120 µg) VR647, 25 breaths (240 µg) VR647, 0.5 mg budesonide, 1 mg budesonide, 5 breaths (30 µg) VR647.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 3, Arm A of single-dose, 4-treatment, 4-period crossover (Other): Subjects received the following treatments in Periods 1 to 4 in a crossover fashion: 15 breaths (120 µg) VR647 via mouthpiece, 15 breaths (120 µg) VR647 via facemask, 0.5 mg budesonide via mouthpiece, 0.5 mg budesonide via facemask.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 3, Arm B of single-dose, 4-treatment, 4-period crossover (Other): Subjects received the following treatments in Periods 1 to 4 in a crossover fashion: 15 breaths (120 µg) VR647 via facemask, 0.5 mg budesonide via mouthpiece, 0.5 mg budesonide via facemask, 15 breaths (120 µg) VR647 via mouthpiece.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 3, Arm C of single-dose, 4-treatment, 4-period crossover (Other): Subjects received the following treatments in Periods 1 to 4 in a crossover fashion: 0.5 mg budesonide via mouthpiece, 0.5 mg budesonide via facemask, 15 breaths (120 µg) VR647 via mouthpiece, 15 breaths (120 µg) VR647 via facemask.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask
- Part 3, Arm D of single-dose, 4-treatment, 4-period crossover (Other): Subjects received the following treatments in Periods 1 to 4 in a crossover fashion: 0.5 mg budesonide via facemask, 15 breaths (120 µg) VR647 via mouthpiece, 15 breaths (120 µg) VR647 via facemask, 0.5 mg budesonide via mouthpiece.
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece; Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece; Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask

INTERVENTIONS:
Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with mouthpiece — The VR647 Inhalation System consists of the AKITA JET control unit that has an inspiration flow rate of 12 L/min, an AKITA JET nebulizer handset, a mouthpiece and dose-specific VR647 Smart Cards designed specifically for this trial.
  Arms: Part 1, Arm A of single-dose, 6-treatment, 6-period crossover; Part 1, Arm B of single-dose, 6-treatment, 6-period crossover; Part 1, Arm C of single-dose, 6-treatment, 6-period crossover; Part 1, Arm D of single-dose, 6-treatment, 6-period crossover; Part 1, Arm E of single-dose, 6-treatment, 6-period crossover; Part 1, Arm F of single-dose, 6-treatment, 6-period crossover; Part 3, Arm A of single-dose, 4-treatment, 4-period crossover; Part 3, Arm B of single-dose, 4-treatment, 4-period crossover; Part 3, Arm C of single-dose, 4-treatment, 4-period crossover; Part 3, Arm D of single-dose, 4-treatment, 4-period crossover
Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System (AKITA JET) with facemask — The VR647 Inhalation System consists of the AKITA JET control unit that has an inspiration flow rate of 12 L/min, an AKITA JET nebulizer handset, a facemask and dose-specific VR647 Smart Cards designed specifically for this trial.
  Arms: Part 2, Arm A of single-dose, 6-treatment, 6-period crossover; Part 2, Arm B of single-dose, 6-treatment, 6-period crossover; Part 2, Arm C of single-dose, 6-treatment, 6-period crossover; Part 2, Arm D of single-dose, 6-treatment, 6-period crossover; Part 2, Arm E of single-dose, 6-treatment, 6-period crossover; Part 2, Arm F of single-dose, 6-treatment, 6-period crossover; Part 3, Arm A of single-dose, 4-treatment, 4-period crossover; Part 3, Arm B of single-dose, 4-treatment, 4-period crossover; Part 3, Arm C of single-dose, 4-treatment, 4-period crossover; Part 3, Arm D of single-dose, 4-treatment, 4-period crossover
Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece — Commercial Pulmicort Respules (budesonide inhalation suspension 1 mg/2 mL) will be delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece operated to sputtering.
  Arms: Part 1, Arm A of single-dose, 6-treatment, 6-period crossover; Part 1, Arm B of single-dose, 6-treatment, 6-period crossover; Part 1, Arm C of single-dose, 6-treatment, 6-period crossover; Part 1, Arm D of single-dose, 6-treatment, 6-period crossover; Part 1, Arm E of single-dose, 6-treatment, 6-period crossover; Part 1, Arm F of single-dose, 6-treatment, 6-period crossover
Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask — Commercial Pulmicort Respules (budesonide inhalation suspension 1 mg/2 mL) will be delivered by a conventional jet nebulizer (PARI VIOS) with facemask operated to sputtering.
  Arms: Part 2, Arm A of single-dose, 6-treatment, 6-period crossover; Part 2, Arm B of single-dose, 6-treatment, 6-period crossover; Part 2, Arm C of single-dose, 6-treatment, 6-period crossover; Part 2, Arm D of single-dose, 6-treatment, 6-period crossover; Part 2, Arm E of single-dose, 6-treatment, 6-period crossover; Part 2, Arm F of single-dose, 6-treatment, 6-period crossover
Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece — Commercial Pulmicort Respules (budesonide inhalation suspension 0.5 mg/2 mL) will be delivered by a conventional jet nebulizer (PARI VIOS) with mouthpiece operated to sputtering.
  Arms: Part 1, Arm A of single-dose, 6-treatment, 6-period crossover; Part 1, Arm B of single-dose, 6-treatment, 6-period crossover; Part 1, Arm C of single-dose, 6-treatment, 6-period crossover; Part 1, Arm D of single-dose, 6-treatment, 6-period crossover; Part 1, Arm E of single-dose, 6-treatment, 6-period crossover; Part 1, Arm F of single-dose, 6-treatment, 6-period crossover; Part 3, Arm A of single-dose, 4-treatment, 4-period crossover; Part 3, Arm B of single-dose, 4-treatment, 4-period crossover; Part 3, Arm C of single-dose, 4-treatment, 4-period crossover; Part 3, Arm D of single-dose, 4-treatment, 4-period crossover
Combination Product: 0.5 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer (PARI VIOS) with facemask — Commercial Pulmicort Respules (budesonide inhalation suspension 0.5 mg/2 mL) will be delivered by a conventional jet nebulizer (PARI VIOS) with facemask operated to sputtering.
  Arms: Part 2, Arm A of single-dose, 6-treatment, 6-period crossover; Part 2, Arm B of single-dose, 6-treatment, 6-period crossover; Part 2, Arm C of single-dose, 6-treatment, 6-period crossover; Part 2, Arm D of single-dose, 6-treatment, 6-period crossover; Part 2, Arm E of single-dose, 6-treatment, 6-period crossover; Part 2, Arm F of single-dose, 6-treatment, 6-period crossover; Part 3, Arm A of single-dose, 4-treatment, 4-period crossover; Part 3, Arm B of single-dose, 4-treatment, 4-period crossover; Part 3, Arm C of single-dose, 4-treatment, 4-period crossover; Part 3, Arm D of single-dose, 4-treatment, 4-period crossover

SUMMARY:
This is a three part, randomized, open-label, crossover, Phase 1 trial in adults. Parts 1 and 2 will enroll healthy male and female subjects. Part 3 will enroll subjects with mild asthma. This study will assess the pharmacokinetics, safety and tolerability of single doses of budesonide delivered by VR647 Inhalation System (AKITA® JET) with mouthpiece or face mask to single doses of budesonide delivered by a conventional jet nebulizer (PARI VIOS®) with mouthpiece or face mask.

DETAILED DESCRIPTION:
For all parts of the study, subjects in the VR647 group will receive VR647 Inhalation Suspension delivered by the VR647 Inhalation System (AKITA JET) with either a mouthpiece or a facemask. Similarly, for all parts of the study, subjects in the comparator group will receive approved doses of budesonide (Pulmicort Respules®) delivered by a conventional jet nebulizer (PARI VIOS) with either a mouthpiece or a facemask.

Part 1:

Subjects who fulfill the enrollment criteria will progress to a comparative single dose, 6-treatment, 6-period crossover trial. Subjects will receive 4 dose levels of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (AKITA JET) (5, 10, 15 and 25 breaths, with targeted doses of 30, 60, 120 and 240 µg) and 2 dose levels of budesonide delivered by a conventional jet nebulizer (PARI VIOS) (0.5 and 1 mg). There will be a Washout Period between each dose of approximately 48 hours. Each subject will be randomized to treatment.

Part 2:

Following an approximate 7-day washout, the same cohort of subjects from Part 1 will progress to a comparative single dose, 6-treatment, 6-period crossover trial. There will be a Washout Period between each dose of approximately 48 hours. Each subject will be randomized to treatment in a 6-way crossover.

Part 3:

Subjects with mild asthma who fulfill the enrollment criteria (including those criteria specific to Part 3) will progress to a comparative single dose, 4-treatment, 4-period crossover trial conducted at a separate clinic from Parts 1 and 2. There will be a Washout Period between each dose of approximately 48 hours. This part of the trial can start before completion of Parts 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject
* Female subjects must have a negative pregnancy test at the Screening and Day -1 Visits (prior to dosing), must be using a reliable form of contraception throughout the trial, or must be of non-childbearing potential as follows:

  * Be post-menopausal (their last menstrual period was at least 12 months ago), and have a serum follicle-stimulating hormone (FSH) level consistent with postmenopausal status as determined by the investigator, or
  * Have undergone a hysterectomy, a bilateral oophorectomy or a bilateral salpingectomy
* Aged 18 to 55 years
* Hemoglobin level of ≥11.5 g/dL for females and ≥13.0 g/dL for males
* Weigh at least 50 kg, and body mass index (Quetelet index) in the range 18.0-32.0 kg/m2, inclusive
* Forced expiratory volume in 1 second (FEV1) of more than 1.69 L at the Screening Visit
* Ability to comprehend the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial
* Give written consent to participate after reading the consent form, and after having the opportunity to discuss the trial with the investigator or his/her delegate

Additional Inclusion Criteria for Part 3:

* Documented clinical history of mild asthma (mild as defined by the National Asthma Evaluation and Prevention Program (NAEPP) guidelines) for at least 6 months before the Screening Visit, but otherwise healthy
* FEV1 reversibility (increase of at least 12% and 200 mL in absolute FEV1 from pre bronchodilator value within 15±5 minutes post bronchodilator) at the Screening Visit or during past 12 months
* Values for FEV1 of at least 80% of predicted value and normal FEV1/forced vital capacity (FVC; as defined by NAEPP guidelines). Assessment should be performed without treatment with β2-agonists. If a subject's FEV1 is outside that range at the Screening Visit, the test may be repeated once on another day during the Screening Period

Exclusion Criteria:

* Clinically relevant abnormal medical history, physical findings, ECG, or laboratory values at the screening assessment that could interfere with the objectives of the trial or the safety of the subject (excluding mild asthma in Part 3)
* Subjects who have impaired cardiovascular, endocrine, autoimmune, metabolic, neurological, renal, respiratory (excluding mild asthma in Part 3), gastrointestinal, hepatic, hematological or any other system abnormalities
* Respiratory tract infection within 4 weeks before the Screening Visit
* History of surgery or medical intervention within 6 weeks before the Screening Visit, or planned surgery or medical intervention, that could interfere with the objectives of the trial or the safety of the subject
* Regular treatment (more than 1 month duration) with oral or parenteral corticosteroids in the last year prior to the Screening Visit
* Use of the following prescription medications within 28 days prior to the first dose:

  * corticosteroids by any route, androgenic steroids (e.g., testosterone), ritonavir and similar drugs for HIV prophylaxis, ketoconazole, itraconazole or similar azole anti-fungal drugs and macrolide antibiotics (e.g., erythromycin)
* Presence or history of severe adverse reaction to any drug, or sensitivity to components of the trial medication
* Use of a prescription or over-the-counter medicine, nutritional and vitamin supplements, with the exception of acetaminophen and hormonal contraceptives, during the 7 days before the first dose of trial medication. For Part 3 only, inhaled short-acting β2-agonists in addition to acetaminophen and hormonal contraceptives are permitted
* Participation in another clinical trial of a new chemical entity, new device, or a prescription medicine within the 3 months before dosing, or participation within 5 half-lives of receiving an experimental drug (whichever is longer)
* Presence or history of drug or alcohol abuse, or intake of more than 21 units (14 units for women) of alcohol weekly
* Evidence of drug abuse on urine testing, or a positive test for alcohol
* Current smoker; or ex-smokers who (a) gave up less than 1 year ago, or (b) who have a history of more than 10 pack years. A pack year is calculated as the number of cigarettes per day multiplied by number of years smoked divided by 20
* Blood pressure and heart rate at the screening examination outside the ranges 90-140 mmHg systolic, 40-90 mm Hg diastolic, heart rate 40-100 beats/min
* Loss of more than 400 mL blood, e.g., as a blood donor, or donation of blood products, during the 3 months before the Screening Visit
* Positive test for hepatitis B, hepatitis C, or HIV
* History of, or latent, tuberculosis (TB) infection
* Evidence of any other clinically significant infection, including bacterial or viral infections
* Possibility that the subject will not cooperate with the requirements of the protocol, including effective use of the nebulizer
* Employee of the investigational site or the Sponsor, who is directly involved in the trial, or a family member of such a person

Additional Exclusion Criteria for Part 3:

* Any life-threatening asthmatic episode in the past
* Asthmatic episode or respiratory tract infection requiring systemic steroid treatment or hospitalization 3 months prior to the Screening Visit
* Use of inhaled short-acting β2-agonists for > 2 days/week for symptom relief during 28 days prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
AUClast (area under the plasma concentration-time curve, from time 0 to the time of the last measurable concentration). | pre-dose and at 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after start of nebulization for Parts 1, 2 and 3
  AUClast (area under the plasma concentration-time curve, from time 0 to the time of the last measurable concentration) compared for single doses of VR647 delivered by VR647 Inhalation System (AKITA JET) with single doses of budesonide delivered by a conventional jet nebulizer (PARI VIOS) via a mouthpiece in healthy volunteers, via a facemask in healthy volunteers, and via either a mouthpiece or a facemask in adult subjects with mild asthma.
AUCinf (area under the plasma concentration-time curve, from time 0 extrapolated to infinity). | pre-dose and at 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after start of nebulization for Parts 1, 2 and 3
  AUCinf (area under the plasma concentration-time curve, from time 0 extrapolated to infinity) compared for single doses of VR647 delivered by VR647 Inhalation System (AKITA JET) with single doses of budesonide delivered by a conventional jet nebulizer (PARI VIOS) via a mouthpiece in healthy volunteers, via a facemask in healthy volunteers, and via either a mouthpiece or a facemask in adult subjects with mild asthma.
Cmax (maximum observed concentration). | pre-dose and at 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after start of nebulization for Parts 1, 2 and 3
  Cmax (maximum observed concentration) compared for single doses of VR647 delivered by VR647 Inhalation System (AKITA JET) with single doses of budesonide delivered by a conventional jet nebulizer (PARI VIOS) via a mouthpiece in healthy volunteers, via a facemask in healthy volunteers, and via either a mouthpiece or a facemask in adult subjects with mild asthma.
Tmax (time to reach Cmax). | pre-dose and at 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after start of nebulization for Parts 1, 2 and 3
  Tmax (time to reach Cmax) compared for single doses of VR647 delivered by VR647 Inhalation System (AKITA JET) with single doses of budesonide delivered by a conventional jet nebulizer (PARI VIOS) via a mouthpiece in healthy volunteers, via a facemask in healthy volunteers, and via either a mouthpiece or a facemask in adult subjects with mild asthma.
T1/2 (apparent first-order terminal elimination half-life). | pre-dose and at 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after start of nebulization for Parts 1, 2 and 3
  T1/2 (apparent first-order terminal elimination half-life) compared for single doses of VR647 delivered by VR647 Inhalation System (AKITA JET) with single doses of budesonide delivered by a conventional jet nebulizer (PARI VIOS) via a mouthpiece in healthy volunteers, via a facemask in healthy volunteers, and via either a mouthpiece or a facemask in adult subjects with mild asthma.

SECONDARY OUTCOMES:
Number of adverse events (AEs) and serious adverse events (SAEs). | Part 1 and Part 2: approximately 64 days; Part 3: approximately 42 days
  Adverse events occurring from the time of the subject giving informed consent until Follow-up/early discontinuation.
Number of adverse device effects (ADEs) and serious adverse device effects (SADEs). | Part 1 and Part 2: approximately 64 days; Part 3: approximately 42 days
  Adverse device effects occurring from the time of the subject giving informed consent until the Follow up/early discontinuation.
Subjects with use of concomitant medications. | Part 1 and Part 2: approximately 64 days; Part 3: approximately 42 days
  Concomitant medication use will be collected and coded using the World Health Organization Drug Dictionary.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Burgess, MD, Study Director — Vectura Ltd
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California